CLINICAL TRIAL: NCT02659254
Title: A First-in-Man Study of the Firesorb Sirolimus Target Eluting Bioresorbable Vascular Scaffold in Patients With Coronary Artery Disease: FUTURE-I
Brief Title: A First-in-Man Study of the Firesorb BVS (FUTURE-I)
Acronym: FUTURE-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai MicroPort Medical (Group) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MicroPort_Firesorb_FIM
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease
Keywords: Drug-Eluting Stents,Absorbable Implants,Stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Firesorb Implantation (Experimental): Implantation of the Sirolimus Target Eluting Bioresorbable Vascular Scaffold （Firesorb）in patients with coronary artery lesions.
  Interventions: Device: Sirolimus Target Eluting Bioresorbable Vascular Scaffold

INTERVENTIONS:
Device: Sirolimus Target Eluting Bioresorbable Vascular Scaffold — Implantation of the Sirolimus Target Eluting Bioresorbable Vascular Scaffold
  Other Names: Firesorb

SUMMARY:
This study is a small scale pilot trial for Sirolimus Target Eluting Bioresorbable Vascular Scaffold (Firesorb) in Patients with Coronary Artery Disease for the first time. The goal is to access the preliminary safety and efficacy of Firesorb implantation in the human body, and to provide evidence for subsequent large-scale, multi-center, randomized controlled clinical trials. Then provide the basis for the formal application of the product in China.

DETAILED DESCRIPTION:
This study is a prospective, single-center clinical trial. The investigator design to recruit 45 subjects. After implanting the Sirolimus Target Eluting Bioresorbable Vascular Scaffold (Firesorb) successfully, all the subjects will be randomly assigned to queue 1 (n=30) and queue 2 (n=15). The clinical follow-up will be performed in all subjects at 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after scaffold implantation. Angiographic,IVUS and OCT follow-up will be performed at 6 months and 2 years after scaffold implantation in queue 1; angiographic,IVUS and OCT follow-up will be performed at 1 year and 3 years after scaffold implantation in queue 2. The primary endpoint of the study is target lesion failure (TLF) at 30 days after scaffold implantation, the secondary endpoints are series of imaging outcomes, for evaluation of feasibility and preliminary safety and efficacy of the product.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years of age, males or non-pregnant females;
2. With silent ischemia evidence, patients with stable or unstable angina, or in patients with old myocardial infarction;
3. Total number of target lesion is 1;
4. Target lesion length ≤ 25mm (Visual); target lesion diameter between 3.0mm to 3.5mm;
5. Visual assessment of target lesion diameter stenosis ≥ 70%,TIMI blood flow≥1;
6. Each target lesion may be covered by a single stent;
7. Patients with indications for coronary artery bypass graft surgery;
8. To understand the purpose of testing, voluntary and informed consent, patients undergoing invasive imaging follow-up.

Exclusion Criteria:

1. Within 1 week of any acute myocardial infarction or myocardial enzymes did not return to normal;
2. Implantation of stent in target vessel within 1 year , patients with planned intervention again within six months;
3. Severe congestive heart failure (NYHA class III and above) ,left ventricular ejection fraction or <40% (ultrasound or left ventricular angiography);
4. Preoperative renal function serum creatinine >2.0mg/DL; receiving hemodialysis;
5. Bleeding, active gastrointestinal ulcers, brain hemorrhage or subarachnoid hemorrhage and half year history of ischemic stroke, antiplatelet agents and would not allow an anticoagulant therapy contraindications patients undergoing antithrombotic therapy;
6. Aspirin, clopidogrel, heparin, contrast agent, poly lactic acid polymer and rapamycin allergies;
7. The patient's life expectancy is less than 12 months;
8. Top participated in other drug or medical device and does not meet the primary study endpoint in clinical trials time frame;
9. Researchers determine patient compliance is poor, unable to complete the study in accordance with the requirements;
10. Heart transplantation patients;
11. The unstable arrhythmia, such as high risk ventricular extrasystole and ventricular tachycardia;
12. Cancer need chemotherapy;
13. Immunosuppression and autoimmune diseases, planned or undergoing immunosuppressive therapy;
14. Planning or being receiving long-term anticoagulant therapy, such as heparin, warfarin, etc;
15. Within six months for elective surgery requires stopping aspirin, Clopidogrel patients;
16. Blood test prompted platelet counts of less than 100x10E9/L or greater than 700x10E9/L, white blood cells than 3x10E9/L; known or suspected liver disease (such as hepatitis);
17. Peripheral vascular disease, 6F catheter is not available.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Device-oriented composite endpoints (Target Lesion Failure) | 1 month after index procedure
  Target Lesion Failure is defined as the composited endpoints of cardiac death,target vessel myocardial infarction and clinical driven-target lesion revascularization.

SECONDARY OUTCOMES:
Target Lesion Failure | 6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Target Lesion Failure is defined as the composited endpoints of cardiac death,target vessel myocardial infarction and clinical driven-target lesion revascularization.
Patient-oriented clinical composite endpoint (PoCE) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Patient-oriented clinical composite endpoint is defined as all cause death, all myocardial infarction, and any revascularization.
Device Success | From the start of index procedure to end of index procedure
  Successful delivery and deployment of the assigned scaffold/stent at the intended target lesion and successful withdrawal of the delivery system with attainment of final in-scaffold/stent residual stenosis of less than 30% by visual.
Procedural Success | At time of procedure up to 7 days in hospital
  Achievement of final in-scaffold/stent residual stenosis of less than 30% by visual estimation with successful delivery and deployment of at least one assigned scaffold/stent at the intended target lesion and successful withdrawal of the delivery system for the target lesion without the occurrence of cardiac death, target vessel MI or repeat TLR.
Scaffold Thrombosis/Stent Thrombosis (per ARC definition) | 1 month,6 months,1 year,2 years,3 years,4 years and 5 years after index procedure
  Timing (acute, sub-acute, late and very late) Evidence (definite and probable)
In-device, in-segment, proximal and distal minimum lumen diameter (MLD) | 6 months,1 year,2 years and 3 years after index procedure
  Angiographic endpoint.
In-device, in-segment, proximal and distal % diameter stenosis (DS) | 6 months,1 year,2 years and 3 years after index procedure
  Angiographic endpoint.
In-device, in-segment, proximal and distal angiographic binary restenosis (ABR) | 6 months,1 year,2 years and 3 years after index procedure
  Angiographic endpoint.
In-device, in-segment,proximal and distal late lumen loss (LLL) | 6 months,1 year,2 years and 3 years after index procedur
  Angiographic endpoint.
Vasomotion | 6 months,1 year,2 years and 3 years after index procedure
  The changes in average lumen diameter before and after intracoronary nitroglycerin.

OTHER OUTCOMES:
Descriptive analysis of morphometric, lesion composition and scaffold strut data obtained with OCT | Immediate,6 months,1 year,2 years and 3 years after index procedure
  OCT endpoint.
Descriptive analysis of vascular and scaffold morphology obtained with IVUS | 6 months,1 year,2 years and 3 years after index procedure
  IVUS endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, MD, Principal Investigator — Fu Wai Hospital & National Center for Cardiovascular Diseases in China
Locations (1):
- Fu Wai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided